CLINICAL TRIAL: NCT06826547
Title: Optimization of Basal Insulin During Ramadan Fasting in Type 2 Diabetic Patients: Comparison Between DAR Recommendations and the Carbohydrate Fasting Test & Metabolic and Inflammatory Consequences
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Collaborators: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Chayma Bel Hadj Sliman, Clinical professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE001
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2 Treated with Insulin; Fasting, Intermittent; Ramadan Fasting; Inflammatory Markers
MeSH Terms: conditions — Diabetes Mellitus; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAR Group (Active Comparator): The basal insulin doses will be adjusted in accordance with the recommendations published by DAR in 2021 for diabetic patients during Ramadan.
  Interventions: Drug: Adjustment of insulin doses DAR
- CFT Group (Active Comparator): The basal insulin doses will be adjusted after a carbohydrate fasting test to assess individual insulin needs during fasting periods.
  Interventions: Drug: Adjustment of insulin doses CFT

INTERVENTIONS:
Drug: Adjustment of insulin doses DAR — Patients will be hospitalized at La Rabta Hospital from February 15 to February 28, 2025 for clinical (weight, BP, SF-12), biological (HbA1c, lipid profile) assessments and inflammatory markers (Interleukin 6 and TNF alfa) DAR Group: Insulin will be adjusted per DAR 2021 guidelines. Patients will track insulin doses, glycemic cycles, hypoglycemia episodes, fasting interruptions, and hospital visits in a dedicated log. They will receive weekly calls for insulin adjustments and continuous support.
  During the last week of Ramadan, clinical and biological data including inflammatory markers will be collected. Two months post-Ramadan, HbA1c, fasting glucose, and lipid profile will be reassessed to evaluate glycemic control.
  Arms: DAR Group
Drug: Adjustment of insulin doses CFT — Patients will be hospitalized at La Rabta Hospital from February 15 to February 28, 2025 for clinical (weight, BP, SF-12) and biological (HbA1c, lipid profile) assessments and inflammatory markers (Interleukin 6 and TNF alfa) .
  CFT Group: Insulin adjusted after a Carbohydrate Fasting Test. Patients will track insulin doses, glycemic cycles, hypoglycemia episodes, fasting interruptions, and hospital visits in a dedicated log. They will receive weekly calls for insulin adjustments and continuous support.
  During the last week of Ramadan, clinical and biological data including inflammatory markers will be collected. Two months post-Ramadan, HbA1c, fasting glucose, and lipid profile will be reassessed to evaluate glycemic control.
  Arms: CFT Group

SUMMARY:
Ramadan, a fasting period observed by many Muslim patients, poses a significant challenge for glycemic management in diabetics. During this month, abstinence from food, water, and medication from dawn to dusk leads to significant glycemic fluctuations. Inadequate insulin dose management can cause acute complications such as hypoglycemia, hyperglycemia, ketosis, or hyperosmolar states. In 2021, the Diabetes and Ramadan (DAR) guidelines provided recommendations for adjusting insulin doses, taking into account changes in circadian rhythms and patients' dietary habits. However, these standardized recommendations may not be suitable for everyone. A personalized alternative, the Carbohydrate Fasting Test (CFT), allows for the assessment of individual basal insulin needs through a controlled fast excluding carbohydrates for 24 hours. Comparing these two approaches could provide valuable insights into their relative effectiveness, particularly in terms of safety and quality of life for patients.

Moreover, diabetes can be influenced by fasting, with potentially beneficial effects on inflammation and metabolism.

This study aims to determine which of these two methods optimizes glycemic control and to assess the variations of inflammation markers before and after Ramadan fasting. The results could be integrated into future clinical practices to improve diabetes management during Ramadan. We aim to compare the effectiveness and safety of basal insulin dose adjustments according to DAR 2021 guidelines versus the Carbohydrate Fasting Test (CFT) and to analyze the impact on the quality of life of diabetic patients. This is a prospective, longitudinal, randomized, interventional study including 60 Type 2 diabetic patients, aged 18 to 70 years old, on insulin therapy for at least 6 months. All participants intend to fast during Ramadan and are at low to moderate risk according to the IDF-DAR score (≤6).

Eligible patients will be randomly assigned into two groups:

DAR Group: Insulin dose adjustments according to DAR 2021 recommendations. CFT Group: Personalized insulin adjustments based on a Carbohydrate Fasting Test conducted before Ramadan.

Protocol:

Initial assessment will be Clinical ( Weight, BMI, blood pressure) and biological (Fasting glucose, HbA1c, fructosamine and inflammatory markers ( Interleukin 6 and TNF alfa)).

During Ramadan, weekly glycemic monitoring will be conducted to track blood sugar levels. Any complications will be recorded, and insulin dose adjustments will be made remotely if necessary to ensure optimal glycemic control.

In the last week of Ramadan, a final clinical assessment will be performed, including measurements of weight, BMI, and blood pressure. A biological assessment will also be conducted to measure fructosamine levels and inflammatory markers ( Interleukin 6 and TNF alfa).

Two months after Ramadan, fasting glucose and HbA1c levels will be re-evaluated to assess long-term glycemic control. The study will also analyze the impact on glycemic regulation, anthropometric parameters, and overall quality of life using the SF-12 questionnaire.

In conclusion, this project aims to identify the most effective method for adjusting basal insulin doses during Ramadan, contributing to optimal Type 2 diabetes management and to assess the variations of inflammation markers before and after Ramadan fasting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years with Type 2 diabetes on a basal insulin regimen (NPH, Detemir, or Glargine) with or without 1 to 2 boluses of rapid-acting insulin.
* Diabetes duration of at least 2 years and insulin therapy for at least 6 months.
* Patients wishing to fast during Ramadan and having provided informed consent.
* Low risk of complications according to the IDF-DAR 2021 risk score or moderate risk for patients who insist on fasting.

Non-Inclusion Criteria:

* High-risk patients according to IDF-DAR 2021 score >6, including those with:
* Severe renal impairment
* Cognitive dysfunction or frailty
* Unrecognized hypoglycemia
* Unstable cardiovascular disease
* Pregnancy
* Type 1 diabetes
* Type 2 diabetes patients on sulfonylureas or related medications

Exclusion Criteria:

* Patients who did not follow the study protocol regarding insulin dose adjustments and capillary blood glucose (CBG) self-monitoring.
* Fasting discontinuation without medical advice.
* Severe complications requiring fasting cessation.
* Patients who withdrew their informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
fructosamine levels | up to 6 weeks
  Fructosamine variation 15 days before & the last week of Ramadan
Interleukin-6 levels | up to 6 weeks
  variation during the fast of Ramadan 15 dayd before and at the Last week of Ramadan
Hypoglycemia | up to one month
  Frequency of hypoglycemic episodes
glycemic auto-monitoring | up to one month
  Percentage of blood glucose values meeting target levels during the month of Ramadan
HbA1c levels | up to 6 weeks
  HbA1c variation before and after Ramadan 15 days before & 2 months after Ramadan
TNF-alfa levels | up to 6 weeks
  Variation during fasting Ramadan 15 days before and at the Last week of Ramadan

SECONDARY OUTCOMES:
Body mass index | up to 6 weeks
  Body mass index variation : Before and at the Last week of Ramadan
Quality of life of patients | up to 6 weeks
  Quality of life of patients assessed using the Medical Outcomes Study Short-Form General Health Survey (SF-12) questionnaire in its validated Tunisian dialect version.
  Before and at at the last week of Ramadan Higher score means a better quality of life.
waist circumference | up to 6 weeks
  variation of waist circumference: Before and at the Last week of Ramadan
Blood pressure | up to 6 weeks
  Variation of blood pressure : Before and at the Last week of Ramadan

IPD SHARING:
Plan to Share IPD: Undecided